CLINICAL TRIAL: NCT05093049
Title: A Pilot Study of the Renuvion APR System When Used as an Adjunct Procedure In Gynecomastia Surgery
Brief Title: Renuvion APR System When Used as an Adjunct Procedure In Gynecomastia Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apyx Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APX-21-02
Record Dates: First submitted 2021-10-13; First posted 2021-10-26 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Gynecomastia
Keywords: Renuvion; Helium Plasma
MeSH Terms: conditions — Gynecomastia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Gynecomastia Surgery Followed by Renuvion (Active Comparator): Patients receiving gynecomastia correction surgery followed by Renuvion treatment were randomly assigned to the left or the right side of the chest in a split-body randomized design. The gynecomastia surgery and Renuvion APR System use will be as per investigator's standard clinical practice.
  Interventions: Device: Renuvion APR System; Procedure: Gynecomastia Correction Surgery
- Gynecomastia Surgery Only (Active Comparator): Patients receiving gynecomastia correction surgery followed by Renuvion treatment were randomly assigned to the left or the right side of the chest in a split-body randomized design. The gynecomastia surgery will be as per investigator's standard clinical practice.
  Interventions: Procedure: Gynecomastia Correction Surgery

INTERVENTIONS:
Device: Renuvion APR System — The Renuvion APR Handpiece (K191542) is a sterile, single use electrosurgical (monopolar) device intended to be used in conjunction with compatible generators for the percutaneous delivery of radiofrequency energy and/or helium plasma for cutting, coagulation and ablation of soft tissue. The Renuvion APR Handpiece is compatible with the Electrosurgical Generators BVX-200H/P (K170188), and APYX-JS3/RS3 (K192867) owned by Apyx Medical that are indicated for delivery of radiofrequency energy and/or helium gas plasma to cut, coagulate, and ablate soft tissue during open and laparoscopic surgical procedures.
  Arms: Gynecomastia Surgery Followed by Renuvion
Procedure: Gynecomastia Correction Surgery — Gynecomastia correction surgery as per the investigators standard treatment of care utilizing liposuction.

SUMMARY:
This is a prospective, multi-center, single-blinded, randomized study of up to 10 study subjects undergoing bilateral gynecomastia surgery with Renuvion APR System used as an adjunct procedure on one side. The study was conducted at a single investigational center in the United States.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-blinded, randomized study of up to 10 study subjects undergoing bilateral gynecomastia surgery with Renuvion APR System used as an adjunct procedure on one side. The study was conducted at a single investigational center in the United States.

At baseline, the grade of gynecomastia was recorded by side, male chest measurements will be taken, and pre-surgery photographs taken in the frontal, lateral, and oblique views.

The gynecomastia surgery and Renuvion APR System use were as per investigator's standard clinical practice. During the procedure, fat transfer and treatment of the lateral chest and/or axilla was not allowed. The Renuvion APR System was used on one side only. The Renuvion treated side was randomized and the patient was blinded as to which side of the chest received Renuvion. Procedure data and adverse events were captured. Endermology was not allowed post-procedure. Post-procedure compression was used for 2-3 weeks with a standard compression vest for all subjects.

Follow-up images, grade of gynecomastia, and male chest measurements were taken at D30/D90/D180.

All images were assessed for correct identification of Renuvion-treated side by blinded Independent Photographic Reviewers (IPR) following the D180 visit.

Following study participation, the subject was offered an optional balancing treatment to the side not previously treated with Renuvion.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects, ages 18 - 75 years old.
2. ASA Physical Status Classification System Class I and Class II subjects.
3. Clinical diagnosis of primary or secondary Gynecomastia.
4. Gynecomastia Rohrich Grade IIA or higher.
5. Symmetrical gynecomastia Rohrich grades.
6. Symmetrical chest measurements (no more than 3% variance between sides).
7. Scheduled for Gynecomastia surgery.
8. Willing to have Renuvion APR System as an adjunct procedure on one side understanding that an optional balancing procedure may be provided post-study exit.
9. Understands and accepts the obligation not to undergo any other procedures or treatments in the areas to be treated during study participation.
10. Absence of physical conditions unacceptable to the investigator.
11. Willing and able to comply with protocol requirements, including study-required images/photos, assessments/measurements, and returning for follow-up visits.
12. Willing to release rights for the use of study photos, including in publication.
13. Able to read, understand, sign, and date the informed consent.

Exclusion Criteria:

1. Subjects without clinical diagnosis of primary Gynecomastia and/or a clinical diagnosis of gynecomastia with secondary causes such as medications, drugs, or testicular tumors.
2. Subjects presenting with ASA Physical Status Classification System Classes III or higher.
3. Gynecomastia Rohrich Grade I.
4. Non-symmetrical gynecomastia Rohrich grades.
5. Non-symmetrical chest measurements (more than 3% variance between sides).
6. Previous treatment or surgery in the breast area.
7. Active systemic or local skin disease that may alter wound healing.
8. Significant or uncontrolled medical condition that in the opinion of the investigator participation in the study may compromise the patient's health.
9. History of autoimmune disease (excluding Hashimoto's thyroiditis).
10. Known susceptibility to keloid formation or hypertrophic scarring.
11. Cancerous or pre-cancerous lesions in the area to be treated.
12. Possesses a surgically implanted electronic device (i.e. pacemaker).
13. Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years.
14. Use of endermology post-procedure for the duration of the study.
15. Participation in any other investigational study within 30 days prior to consent and throughout study participation.
16. Subject who, in the opinion of the investigator, is not an appropriate candidate for the study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Ruff, MD, Principal Investigator — West End Plastic Surgery
Locations (1):
- West End Plastic Surgery, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from a single site in the United States.
Pre-assignment Details: All ten subjects in need of gynecomastia correction surgery were treated in a bilateral randomized design. One side of the chest received gynecomastia surgery. The other side received gynecomastia surgery followed by treatment with Renuvion.
Units Other Than Participants: Treatment Modality
Groups:
- Gynecomastia Surgery Only: Patients receiving gynecomastia correction surgery were randomly assigned to the left or the right side of the chest in a split-body randomized design.
- Gynecomastia Surgery Followed by Renuvion: Patients receiving gynecomastia correction surgery followed by Renuvion treatment were randomly assigned to the left or the right side of the chest in a split-body randomized design.
Period: Overall Study
Arm/Group | Gynecomastia Surgery Only | Gynecomastia Surgery Followed by Renuvion
Started | 10; 10 Treatment Modality | 10; 10 Treatment Modality
Completed (Ten subjects were enrolled in the study and treated bilaterally.) | 10; 10 Treatment Modality | 10; 10 Treatment Modality
Not Completed | 0; 0 Treatment Modality | 0; 0 Treatment Modality

BASELINE CHARACTERISTICS:
Population: Male subjects were enrolled who needed gynecomastia correction surgery.
Groups:
- All Subjects: Total of all reporting groups
Arm/Group | All Subjects
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 41 [19 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
BMI [Mean (Full Range); unit: kg/m^2] | 26.5 [20.6 to 30.8]
Rohrich Classification of Gynecomastia [Count of Participants; unit: Participants] — Grade I (Minimal hypertrophy, <250g of breast tissue, without ptosis) I A: Primarily glandular* I B: Primarily fibrous* Grade II (Moderate hypertrophy, 250-500g of breast tissue, without ptosis) I A: Primarily glandular* I B: Primarily fibrous* Grade III (Severe hypertrophy, >500g of breast tissue, with grade I ptosis Glandular or fibrous*) Grade IV (Severe hypertrophy with grade I or III ptosis) Glandular or fibrous*
  *Fatty and glandular tissue is determined by a pinch test medially, laterally, and beneath the nipple-areola complex
  Participants
    Grade IIA | 8
    Grade IIB | 2

OUTCOME MEASURES:

1. Primary Outcome: Analysis of Bilateral Occurrence of Adverse Events
Description: Analysis of bilateral occurrence of adverse events by study arm.
Time Frame: Through Day 180
Population: Healthy, male adult subjects, ages 18 - 75 years old who meet the inclusion/exclusion criteria.
Measure: Number; unit: Number of Events
Arm/Group | Gynecomastia Surgery Followed by Renuvion | Gynecomastia Surgery Only
Number analyzed (Participants) | 10 | 10
Number of Events
  Number of Expected Treatment Effects | 42 | 38
  Number of Adverse Events | 6 | 7

2. Secondary Outcome: Bilateral Analysis of Change to Soft-Tissue Pinch Thickness of the Upper Pole
Description: A measurement of the soft-tissue pinch thickness of the upper pole, by isolating skin and subcutaneous tissue superior to the breast parenchyma, pinching firmly, and measuring the thickness with a caliper.
Time Frame: Day 30, 90, 180
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Gynecomastia Surgery Followed by Renuvion | Gynecomastia Surgery Only
Number analyzed (Participants) | 10 | 10
cm
  Change from Baseline to D30 | -0.29 (0.37) | -0.31 (0.52)
  Change from Baseline to D90 | -0.49 (0.51) | -0.59 (0.51)
  Change from Baseline to D180 | -0.59 (0.53) | -0.72 (0.5)

3. Secondary Outcome: Bilateral Analysis of Change to Soft-Tissue Pinch Thickness at the Inframammary Fold
Description: A measurement of soft-tissue pinch thickness at the inframammary fold by isolating skin and subcutaneous tissue at the inframammary fold, pinching firmly, and measuring the thickness with a caliper.
Time Frame: Day 30, 90, 180
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Gynecomastia Surgery Followed by Renuvion | Gynecomastia Surgery Only
Number analyzed (Participants) | 10 | 10
cm
  Change from Baseline to D30 | -0.11 (.022) | -0.24 (0.29)
  Change from Baseline to D90 | -0.16 (0.27) | -0.28 (0.22)
  Change from Baseline to D180 | -0.17 (0.23) | -0.29 (0.26)

4. Secondary Outcome: Bilateral Analysis of Male Chest Measurements
Description: Measurement of suprasternal notch to nipple, inter-nipple distance, suprasternal notch to nipple plane, midclavicular point to nipple, nipple plane to umbilicus, umbilicus to pubic symphysis, coracoid process to nipple plane, nipple plane to medial epicondyle, and coracoid process to medial epicondyle.
Time Frame: Day 30, 90, 180
Measure: Mean (Full Range); unit: cm
Arm/Group | Gynecomastia Surgery Followed by Renuvion | Gynecomastia Surgery Only
Number analyzed (Participants) | 10 | 10
cm
  Change in Suprasternal Notch to Nipple from Baseline to D30 | -0.1 [-1.0 to 0.5] | 0 [-0.5 to 0.2]
  Change in Suprasternal Notch to Nipple from Baseline to D90 | -0.1 [-1.0 to 1.0] | 0 [-1.0 to 0.5]
  Change in Suprasternal Notch to Nipple from Baseline to D180 | -0.3 [-0.3 to -1.0] | -0.1 [-1.0 to 0.5]
  Change in Internipple Distance from Baseline to D30 | -0.4 [-2.5 to 1.0] | -0.4 [-2.5 to 1.0]
  Change in Internipple Distance from Baseline to D90 | -0.7 [-2.5 to 0] | -0.7 [-2.5 to 0]
  Change in Internipple Distance from Baseline to D180 | -0.8 [-2.0 to 0] | -0.8 [-2.0 to 0]
  Change in Suprasternal Notch to Nipple Plane from Baseline to D30 | -1.8 [-6.0 to 0.5] | -2.0 [-6.5 to 0.5]
  Change in Suprasternal Notch to Nipple Plane from Baseline to D90 | -3.5 [-6.5 to -3.5] | -3.5 [-7.0 to 0]
  Change in Suprasternal Notch to Nipple Plane from Baseline to D180 | -3.4 [-7.0 to -3.4] | -3.5 [-7.5 to -0.5]
  Change in Midclavicular Point to Nipple from Baseline to D30 | 0.1 [-0.5 to 0.5] | 0 [-1.0 to 0.5]
  Change in Midclavicular Point to Nipple from Baseline to D90 | 0.2 [-1.0 to 3.0] | 0.3 [-1.5 to 4.5]
  Change in Midclavicular Point to Nipple from Baseline to D180 | 0.1 [-1.5 to 2.5] | 0.3 [-1.0 to 4.0]
  Change in Nipple Plane to Umbilicus from Baseline to D30 | -0.4 [-1.5 to 0.5] | -0.4 [-1.5 to 0.5]
  Change in Nipple Plane to Umbilicus from Baseline to D90 | -0.4 [-2.0 to 1.0] | -0.4 [-2.0 to 1.0]
  Change in Nipple Plane to Umbilicus from Baseline to D180 | -0.3 [-1.5 to 0.5] | -0.3 [-1.5 to 0.6]
  Change in Umbilicus to Pubic Symphysis from Baseline to D30 | 0 [0 to 0] | 0 [0 to 0]
  Change in Umbilicus to Pubic Symphysis from Baseline to D90 | 0 [0 to 0] | 0 [0 to 0]
  Change in Umbilicus to Pubic Symphysis from Baseline to D180 | 0 [0 to 0] | 0 [0 to 0]
  Change in Coracoid Process to Nipple Plane from Baseline to D30 | 0.1 [-1.0 to 0.5] | -0.1 [-1.0 to 0.5]
  Change in Coracoid Process to Nipple Plane from Baseline to D90 | 0.2 [-1.5 to 1.0] | 0.1 [-1.5 to 1.5]
  Change in Coracoid Process to Nipple Plane from Baseline to D180 | 0.1 [-2.0 to 1.0] | 0.2 [-1.5 to 1.0]
  Change in Nipple Plane to Medial Epicondyle from Baseline to D30 | -0.1 [-1.0 to 1.0] | -0.1 [-1.3 to 1.0]
  Change in Nipple Plane to Medial Epicondyle from Baseline to D90 | -0.2 [-1.0 to 1.5] | -0.3 [-1.5 to 1.5]
  Change in Nipple Plane to Medial Epicondyle from Baseline to D180 | -0.2 [-1.0 to 2.0] | -0.4 [-1.5 to 1.5]
  Change in Coracoid Process to Medial Epicondyle from Baseline to D30 | 0 [0 to 0] | 0 [0 to 0]
  Change in Coracoid Process to Medial Epicondyle from Baseline to D90 | 0 [0 to 0] | 0 [0 to 0]
  Change in Coracoid Process to Medial Epicondyle from Baseline to D180 | 0 [0 to 0] | 0 [0 to 0]

5. Secondary Outcome: Bilateral Analysis of the Amount of Skin Excised During the Procedure by Gynecomastia Grade (Rohrich Classification)
Description: Bilateral measurement of the amount of skin excised during the procedure (if any) by Gynecomastia Grade (Rohrich Classification). Grade I (Minimal hypertrophy, <250g of breast tissue, without ptosis) I A: Primarily glandular* I B: Primarily fibrous* Grade II (Moderate hypertrophy, 250-500g of breast tissue, without ptosis) I A: Primarily glandular* I B: Primarily fibrous* Grade III (Severe hypertrophy, >500g of breast tissue, with grade I ptosis Glandular or fibrous*) Grade IV (Severe hypertrophy with grade I or III ptosis) Glandular or fibrous*
  *Fatty and glandular tissue is determined by a pinch test medially, laterally, and beneath the nipple-areola complex
Time Frame: Procedure
Population: None of the patients in this study had skin excised during treatment, thus none were analyzed for this endpoint which was looking at how much skin was excised by their Gynecomastia Grade. In the case of this study, it was none.
Arm/Group | Gynecomastia Surgery Followed by Renuvion | Gynecomastia Surgery Only
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Gland Tissue Removal by Number of Participants
Description: Bilateral analysis of the number of subjects with gland tissue removed by the during the procedure. The technique utilized for subjects in this study was a mixed surgical technique. The Investigator removed progressive strips of gland in a radial fashion until optimal extraction by palpation was achieved.
Time Frame: Procedure
Measure: Number; unit: participants
Groups:
- Gynecomastia Surgery Followed by Renuvion; Gynecomastia Surgery Only: The gynecomastia surgery and Renuvion APR System were used as per investigator's standard clinical practice. During the procedure, fat transfer and treatment of the lateral chest and/or axilla were not allowed. The Renuvion APR System was used on one side only. The treated side was randomized, and the patient was blinded as to which side of the chest received Renuvion. Procedure data and adverse events were captured. Endermology was not allowed post-procedure. Post-procedure compression was used for 2-3 weeks with a standard compression vest for all subjects.
Arm/Group | Gynecomastia Surgery Followed by Renuvion | Gynecomastia Surgery Only
Number analyzed (Participants) | 10 | 10
participants
  Excision | 2 | 2
  No Excision | 8 | 8

7. Secondary Outcome: Bilateral Physician Global Aesthetic Improvement Scale
Description: The Principal Investigator, sub-investigator or qualified clinician delegated by the principal investigator, will complete a bilateral Physician Global Aesthetic Improvement Scale assessing overall aesthetic improvement in the treatment area. Rating scale: Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse
Time Frame: Day 30, 90, 180
Measure: Count of Participants; unit: Participants
Arm/Group | Gynecomastia Surgery Followed by Renuvion | Gynecomastia Surgery Only
Number analyzed (Participants) | 10 | 10
Participants
  D30: Very Much Improved | 2 | 2
  D30: Much Improved | 5 | 4
  D30: Improved | 2 | 4
  D30: No Change | 1 | 0
  D30: Worse | 0 | 0
  D30: Much Worse | 0 | 0
  D30: Very Much Worse | 0 | 0
  D90: Very Much Improved | 6 | 2
  D90: Much Improved | 2 | 7
  D90: Improved | 2 | 1
  D90: No Change | 0 | 0
  D90: Worse | 0 | 0
  D90: Much Worse | 0 | 0
  D90: Very Much Worse | 0 | 0
  D180: Very Much Improved | 6 | 6
  D180: Much Improved | 4 | 3
  D180: Improved | 0 | 1
  D180: No Change | 0 | 0
  D180: Worse | 0 | 0
  D180: Much Worse | 0 | 0
  D180: Very Much Worse | 0 | 0

8. Secondary Outcome: Bilateral Subject Global Aesthetic Improvement Scale
Description: The subject will complete a bilateral Subject Global Aesthetic Improvement Scale assessing overall aesthetic improvement in the treatment area. Rating scale: Very Much Improved, Much Improved, Improved, No Change, Worse, Much Worse, Very Much Worse
Time Frame: Day 30, 90, 180
Measure: Count of Participants; unit: Participants
Arm/Group | Gynecomastia Surgery Followed by Renuvion | Gynecomastia Surgery Only
Number analyzed (Participants) | 10 | 10
Participants
  D30: Very Much Improved | 4 | 3
  D30: Much Improved | 4 | 4
  D30: Improved | 2 | 3
  D30: No Change | 0 | 0
  D30: Worse | 0 | 0
  D30: Much Worse | 0 | 0
  D30: Very Much Worse | 0 | 0
  D90: Very Much Improved | 4 | 5
  D90: Much Improved | 5 | 5
  D90: Improved | 1 | 0
  D90: No Change | 0 | 0
  D90: Worse | 0 | 0
  D90: Much Worse | 0 | 0
  D90: Very Much Worse | 0 | 0
  D180: Very Much Improved | 5 | 5
  D180: Much Improved | 3 | 4
  D180: Improved | 2 | 1
  D180: No Change | 0 | 0
  D180: Worse | 0 | 0
  D180: Much Worse | 0 | 0
  D180: Very Much Worse | 0 | 0

9. Secondary Outcome: Bilateral Patient Satisfaction Questionnaire
Description: The subject will complete a bilateral Patient Satisfaction Questionnaire for the evaluation of satisfaction for the right side and for the left side. Questions were Yes/No responses.
Time Frame: Day 30, 90, 180
Measure: Count of Participants; unit: Participants
Arm/Group | Gynecomastia Surgery Followed by Renuvion | Gynecomastia Surgery Only
Number analyzed (Participants) | 10 | 10
Participants
  Happy with the results | 9 | 10
  Noted more chest definition | 8 | 8
  Noted improvement in skin texture in the treatment area | 6 | 5
  Noticed a difference in the sides of the chest | 9 | 9
  Believed this side side looked better | 3 | 6
  Requested a balancing procedure | 7 | 7
  Would recommend the procedure to a friend | 9 | 10

10. Secondary Outcome: Correct Identification of Renuvion-treated Side by Blinded Independent Photographic Reviewers
Description: Three experienced, blinded photographic reviewers performed a qualitative analysis/review of pre-treatment and post-treatment sets of images for each subject. Images were provided in a blinded and randomized order. Each blinded reviewer choose which side of the chest was treated with gynecomastia correction surgery followed by Renuvion treatment. Success was the correct identification of treated side of the chest by at least 2 of the 3 reviewers.
Time Frame: Day 180
Measure: Number; unit: Correctly identified side.
Groups:
- All Study Participants: Total of all reporting groups.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
Correctly identified side. | 5

ADVERSE EVENTS:
Time Frame: 180 days
Description: An expected treatment effect was defined as any typical treatment side-effect of Renuvion APR System of mild to moderate severity and lasting up to a typical maximum duration. An adverse event was defined as any new medical problem, or exacerbation of an existing problem, experienced by a subject while enrolled in the study, whether or not it is considered device-related by the investigator.
Groups:
- Liposuction + Renuvion Side of Chest; Liposuction-only Side of the Chest: The gynecomastia surgery and Renuvion APR System were used as per investigator's standard clinical practice. During the procedure, fat transfer and treatment of the lateral chest and/or axilla were not allowed. The Renuvion APR System was used on one side only. The treated side was randomized, and the patient was blinded as to which side of the chest received Renuvion. Procedure data and adverse events were captured. Endermology was not allowed post-procedure. Post-procedure compression was used for 2-3 weeks with a standard compression vest for all subjects.
Arm/Group | Liposuction + Renuvion Side of Chest | Liposuction-only Side of the Chest
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposuction + Renuvion Side of Chest (N=10) | Liposuction-only Side of the Chest (N=10)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Subcutaneous Induration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 2 (2) | 2 (2)
Nausea (General disorders) | 2 (2) | 2 (2)
Surface Paresthesia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations include limited subject numbers, potential variation in subject positioning between visits which can affect measurements, and split body design which due to natural body asymmetry between sides made it challenging to interpret results of the cohorts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT05093049/Prot_000.pdf